CLINICAL TRIAL: NCT03979326
Title: Biomechanical Changes in Young Women During Menstrual Cycle
Brief Title: Biomechanical Changes During Menstrual Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Michalik, Principal Investigator, Medical University of Silesia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: stretching w cyklu
Record Dates: First submitted 2019-02-13; First posted 2019-06-07 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Menstrual Cycle; Passive Stretching; Hamstring Muscles
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young women during various of phases of menstrual cycle. (Experimental): The group of 40 young women will have their hamstring muscle stretched in different phases of the menstrual cycle: follicular, ovulatory and luteal. Static stretching will last 3x 45 seconds with a 15 second break between repetitions. Before and after the intervention a series of tests will be performed.
  Interventions: Procedure: Static stretching

INTERVENTIONS:
Procedure: Static stretching — Static stretching lasting 3 x 45 seconds will be performed in each of the examined women three times in different phases of the menstrual cycle: follicular, ovulatory and luteal. Before and after the intervention, a series of tests assessing the influence of stretching on biomechanical parameters will be carried out

SUMMARY:
The aim of the work is to assess the effect of the menstrual cycle on the biomechanical properties of the muscles. The study will be conducted among young women aged 20-25 with a regular menstrual cycle. During the test, muscle strength and muscle flexibility as well as activation times will be performed. The study will assess the effect of the stretching of the hamstring muscles on the biomechanical properties of the muscles in the different phases of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycle lasting 28 days (+/- 5 days)
* A menstrual cycle that has been present for at least 2 years
* No hormonal contraception
* Lack of pain in the lower spine
* No restriction of mobility in the hip joint

Exclusion Criteria:

* Irregular menstrual cycle
* BMI value below 18.5 and above 25
* Orthopedic disorders in the lower limb
* Neurological disorders
* Normal flexibility of the hamstring muscles

Ages: 20 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Hamstring flexibility | Change measured before and immediately after static stretching during follicular phase of menstrual cycle
  Hamstring flexibility will be assessed using AKE and PKE and SLR tests.
Hamstring flexibility | Change measured before and immediately after static stretching during ovulation phase of menstrual cycle
  Hamstring flexibility will be assessed using AKE and PKE and SLR tests.
Hamstring flexibility | Change measured before and immediately after static stretching during luteal phase of menstrual cycle
  Hamstring flexibility will be assessed using AKE and PKE and SLR tests.
Passive Hamstring flexibility | Change measured before and immediately after static stretching during follicular phase of menstrual cycle
  Hamstring flexibility will be assessed using PKE test
Passive Hamstring flexibility | Change measured before and immediately after static stretching during ovulation phase of menstrual cycle
  Hamstring flexibility will be assessed using PKE test
Passive Hamstring flexibility | Change measured before and immediately after static stretching during luteal phase of menstrual cycle
  Hamstring flexibility will be assessed using PKE test
Active Hamstring flexibility | Change measured before and immediately after static stretching during follicular phase of menstrual cycle
  Hamstring flexibility will be assessed using SLR tests.
Active Hamstring flexibility | Change measured before and immediately after static stretching during ovulation phase of menstrual cycle
  Hamstring flexibility will be assessed using SLR tests.
Active Hamstring flexibility | Change measured before and immediately after static stretching during luteal phase of menstrual cycle
  Hamstring flexibility will be assessed using SLR tests.
Hamstring passive stifness | Change measured before and immediately after static stretching during follicular phase of menstrual cycle
  Hamstring stiffness will be assessed using TDK test. During the test the resistance of the elongated Hamstring muscle is measured. If the resistance value is smaller after the intervention it means that muscle stiffness changed.
Hamstring passive stifness | Change measured before and immediately after static stretching during ovulation phase of menstrual cycle
  Hamstring stiffness will be assessed using TDK test. During the test the resistance of the elongated Hamstring muscle is measured. If the resistance value is smaller after the intervention it means that muscle stiffness changed.
Hamstring passive stifness | Change measured before and immediately after static stretching during luteal phase of menstrual cycle
  Hamstring stiffness will be assessed using TDK test. During the test the resistance of the elongated Hamstring muscle is measured. If the resistance value is smaller after the intervention it means that muscle stiffness changed.
Trunk acivity is assessed using Stabilizer Pressure Biofeedback | Three repetitions with a 30-second break between. The measure is taken during follicular phase of menstrual cycle
  The torso activation scheme is measured during lower and upper limb motions using Chattanooga Stabilizer Pressure Biofeedback.
Trunk acivity is assessed using Stabilizer Pressure Biofeedback | Three repetitions with a 30-second break between. The measure is taken during ovulation phase of menstrual cycle
  The torso activation scheme is measured during lower and upper limb motions using Chattanooga Stabilizer Pressure Biofeedback.
Trunk acivity is assessed using Stabilizer Pressure Biofeedback | Three repetitions with a 30-second break between. The measure is taken during luteal phase of menstrual cycle
  The torso activation scheme is measured during lower and upper limb motions using Chattanooga Stabilizer Pressure Biofeedback.
Hamstring strength is tested using the Micro Fet Handheld Dynamometer. | Change measured before and immediately after static stretching. The measure is taken during follicular phase of menstrual cycle
  Muscle strength of hamstring is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants are asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
Hamstring strength is tested using the Micro Fet Handheld Dynamometer. | Change measured before and immediately after static stretching. The measure is taken during ovulation phase of menstrual cycle
  Muscle strength of hamstring is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants are asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
Hamstring strength is tested using the Micro Fet Handheld Dynamometer. | Change measured before and immediately after static stretching. The measure is taken during luteal phase of menstrual cycle
  Muscle strength of hamstring is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants are asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
Strength of arm flexors and extensors and hip flexors is tested using the Micro Fet Handheld Dynamometer. | Three repetitions for 5-7 seconds with two 30-second intervals . The measure is taken during follicular phase of menstrual cycle
  Muscle strength of arm flexors and extensors and hip flexors is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants are asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
Strength of arm flexors and extensors and hip flexors is tested using the Micro Fet Handheld Dynamometer. | Three repetitions for 5-7 seconds with two 30-second intervals . The measure is taken during ovulation phase of menstrual cycle
  Muscle strength of arm flexors and extensors and hip flexors is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants are asked to press against the Dynamometer with the maximum effort for 5-7 seconds.
Strength of arm flexors and extensors and hip flexors is tested using the Micro Fet Handheld Dynamometer. | Three repetitions for 5-7 seconds with two 30-second intervals . The measure is taken during luteal phase of menstrual cycle
  Muscle strength of arm flexors and extensors and hip flexors is tested. Three repetitions of muscle strength testing are performed with two 30-second intervals. The participants are asked to press against the Dynamometer with the maximum effort for 5-7 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Dąbrowska-Galas, Study Chair — Department of Kinesitherapy and Special Methods, SHS in Katowice, Medical University of Silesia
Locations (1):
- Department of Kinesitherapy and Special Methods, SHS in Katowice, Medical University of Silesia, Katowice, Poland, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study will be available from the corresponding author on reasonable request.